CLINICAL TRIAL: NCT05005000
Title: Autologous Intra-Articular Micro-Fragmented Adipose Transfer for the Treatment of Thumb Carpometacarpal Joint Arthritis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulties getting subjects recruited and enrolled.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-00996
Record Dates: First submitted 2021-08-12; First posted 2021-08-13 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Arthritis
MeSH Terms: conditions — Arthritis | interventions — Triamcinolone Acetonide; Triamcinolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- MFAT (Experimental)
  Interventions: Biological: Micro-Fragmented Adipose Tissue (MFAT)
- Steroid (Control) (Active Comparator)
  Interventions: Drug: Triamcinolone Acetonide 10mg/mL

INTERVENTIONS:
Biological: Micro-Fragmented Adipose Tissue (MFAT) — 1ml of autologous micro-fragmented adipose tissue will be used.
  Arms: MFAT
Drug: Triamcinolone Acetonide 10mg/mL — The control group will receive a 1ml intraarticular injection of triamcinolone acetonide 10mg/ml.
  Other Names: Kenalog-10
  Arms: Steroid (Control)

SUMMARY:
32 patients with Eaton-Glickel stage 2-3 CMC arthritis will be randomized to receive intraarticular MFAT or intraarticular corticosteroid injection. Patients with inflammatory arthritis or prior thumb base trauma or surgery will be excluded. Autologous adipose tissue will be harvested from the outer thigh or lower abdomen using local anesthesia. Tissue will be processed to remove oil and debris in-office using an FDA-approved commercially available device. The processed adipose will be immediately injected into the thumb CMC joint under fluoroscopic guidance. Visual analogue score (VAS), grip/pinch strength, Kapandji range of motion score, thumb disability examination, and QuickDASH score will be assessed pre-procedure and at 2 weeks, 6 weeks, 3 months, 6 months, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old or older; male and female patients
2. Eaton-Glickel stage 2-3 thumb CMC arthritis
3. Failed conservative treatment (i.e. hand therapy, pain medications, splinting)
4. Able to provide informed consent

Exclusion Criteria:

1. Pregnancy/breastfeeding
2. Inflammatory or posttraumatic arthritis
3. Prior thumb base trauma or surgery
4. Evidence of skin infection or soft tissue loss at the thumb CMC joint or adipose harvest site
5. Active local or systemic malignancy
6. Known allergy to any study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05-12 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2023-05-25 (Actual)

PRIMARY OUTCOMES:
Percent Change in Score on Pain Visual Analog Scale (VAS) | Baseline, Month 12
  Pain severity scores will be assessed by use of a visual analog scale (VAS; total range = 0-10; 0 = no pain, 10 = worst pain imaginable)

SECONDARY OUTCOMES:
Change in Score on Thumb Disability Exam (TDX) | Baseline, Month 12
  TDX consists of 20 questions and assess the function of the participant's thumbs over the past week. Each question is scored from 1 (not difficult) to 5 (unable).
  TDX is scored on a scale of 1 to 100, with a higher score indicating a greater degree of disability in the thumb.
Change in Shortened Disabilities of the Arm, Shoulder, and Hand (QuickDASH) Score | Baseline, Month 12
  QuickDASH consists of 11 questions -- the participants are asked to rate their ability to do activities in the last week on a scale of 1 (no difficulty) to 5 (unable). The disability/symptom score is calculated by ((sum of n responses/n)-1)x25, where n is equal to the number of completed responses. The total score ranges from 0 to 250; higher scores indicate greater degree of disability.
Change in Kapandji Range of Motion Score | Baseline, Month 12
  A Kapandji score is used to assess the movement of opposition (being able to touch one's thumb to areas of one's hand). It is vital in hand function and grip. The total score ranges from 1 to 10; a higher score indicates the thumb being able to touch a further area on the hand.

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Hacquebord, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data upon reasonable request. Requests should be directed to Jacques.Hacquebord@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.